CLINICAL TRIAL: NCT04781946
Title: A Pilot Clinical Trial on the Management of Symptomatic Gastric Sleeve Stenosis After Laparoscopic Sleeve Gastrectomy
Brief Title: Management of Symptomatic Gastric Sleeve Stenosis After Laparoscopic Sleeve Gastrectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided not to move forward with the study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00269201
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Gastric Stenosis
Keywords: gastric stenosis; laparoscopic sleeve gastrectomy; bariatric complications; endoscopy
MeSH Terms: interventions — Pyloromyotomy; Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Endoscopic pneumatic balloon dilation (PBD), gastric peroral endoscopic myotomy (G-POEM) and Roux-en-Y gastric bypass (RYGB) will be used for the management of post-LSG GSS using a predefined treatment algorithm.
  Interventions: Procedure: Endoscopic pneumatic balloon dilation; Procedure: Gastric peroral endoscopic myotomy (G-POEM); Procedure: Roux-en-Y gastric bypass (RYGB)

INTERVENTIONS:
Procedure: Endoscopic pneumatic balloon dilation — Using endoscopy, pneumatic balloon dilation may be used to treat stenosis of the gastric sleeve.
Procedure: Gastric peroral endoscopic myotomy (G-POEM) — Gastric per-oral endoscopic myotomy (G-POEM) is a recent innovation offering a minimally invasive endoscopic approach. G-POEM allows for the creation of a tunnel and subsequent myotomy from the gastric cardia to the gastric pylorus.
Procedure: Roux-en-Y gastric bypass (RYGB) — The Roux-en-Y gastric bypass is a type of weight-loss surgery that involves creating a small pouch from the stomach and connecting the newly created pouch directly to the small intestine.

SUMMARY:
The global obesity epidemic has led to increasing popularity of bariatric surgeries and a parallel rise in the prevalence of related complications. Gastric sleeve stenosis (GSS) complicates 0.1-3.9% of cases after Sleeve Gastrectomy (SG) and can result in significant symptoms including nausea, vomiting, epigastric pain, dysphagia, reflux and regurgitation. There is no validated algorithm for the management of GSS, and available literature is retrospective.

The investigators hypothesize that the implementation of a predefined treatment algorithm for management of GSS post SG will effectively and safely manage patients with this condition. This single center, prospective, non-randomized pilot clinical trial to be performed at Johns Hopkins Medical Institutes will describe the efficacy and safety of endoscopic pneumatic balloon dilation (PBD), gastric peroral endoscopic myotomy (G-POEM) and Roux-en-Y gastric bypass (RYGB) for the management of post-LSG GSS using a predefined treatment algorithm. Patients with symptomatic, endoscopically or radiologically confirmed GSS greater than four weeks from laparoscopic sleeve gastrectomy (LSG) who are treatment naïve will be included.

The primary outcome is the rate of clinical success, defined an improvement in symptoms that allowed the patient to avoid further intervention (outside of the predefined treatment algorithm) with a resumption of adequate oral intake and at least 1-point reduction in the Patient Assessment of upper Gastrointestinal Symptoms (PAGI-SYM) questionnaire, at 6 months following last intervention. Secondary outcomes include rates of technical success (completion of planned procedure), procedural success (defined as a 1-point reduction in PAGI-SYM score at 8 weeks following procedure), endoscopic and radiologic resolution of GSS-related findings, percentage of patients maintained off proton pump inhibitor (PPI) therapy, time to recurrence of symptoms post-treatment in patients with recurrence, and rate of adverse events. The expected study population is 30 participants with a study duration of 18 months. This study can potentially validate a treatment algorithm, thereby assisting clinicians to select the most appropriate intervention for the treatment of post-LSG GSS. Moreover, it may help improve outcomes and prevent unnecessary procedures in patients with GSS.

DETAILED DESCRIPTION:
Gastric sleeve stenosis (GSS) can either be mechanical from a short, circumferential stricture (non-helical) or functional secondary to an axial deviation (helical). Helical GSS are believed to be due to asymmetric traction and/or misalignment while stapling, causing a rotated gastric sleeve and functional obstruction to flow. Current treatment options include: endoscopic pneumatic balloon dilation (PBD), endoscopic stenting and revision surgery. Endoscopic balloon dilation demonstrates an overall clinical success rate of 76%[ and usually requires more than one session. However, the optimal size and type of balloon used, as well as the frequency of dilations remains unclear. Additionally, the accessibility and length of the GSS will also impact balloon choice and can occasionally prohibit balloon placement or distension. Endoscopic placement of fully covered self-expanding metal stents (FCSEMS) are effective in 70% of EBD failures. However, FCSEMS have a migration risk of up to 62% in the post-bariatric stricture setting, which may be reduced by suturing. Further, both of these treatment modalities have limited long term success in the setting of helical GSS. Revision surgery, usually a conversion to RYGB is effective in 91% of EBD failures - however can be associated with high adverse event rates. Gastric per-oral endoscopic myotomy (G-POEM) is a recent innovation offering a minimally invasive endoscopic approach. G-POEM allows for the creation of a tunnel and subsequent myotomy from the gastric cardia to the gastric pylorus. Initially developed for the treatment of gastroparesis, case reports have now demonstrated its successful use in post-LSG GSS. A modification to the original technique allows the staple line to be targeted for myotomy, relieving the tortuosity seen in a helical GSS. Case reports and retrospective studies have been supportive of this but there is no prospective data. Currently, there are no clear guidelines on the management of GSS post-LSG and available literature is largely retrospective. Hence, we sought to prospectively evaluated the use of G-POEM for management of patients with symptomatic, endoscopically or radiologically confirmed helical GSS

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms of dysphagia, abdominal pain, nausea, vomiting, heartburn or regurgitation after LSG that do not respond to standard medical therapies, such as proton pump inhibitors, anti-emetics, etc
* Patients with a confirmed sleeve stenosis by contrast study and/or upper endoscopy
* Adult patients aged greater than 18 years old at time of consent
* Patients able to provide written informed consent on the Institutional Review Board/Ethics Committee-approved informed consent form
* Patients willing and able to comply with study requirements for follow up

Exclusion Criteria:

* Presence of concomitant gastric leak or fistula
* Stenosis of non-gastric origin
* History of Roux-en-Y gastric bypass, or duodenal switch
* GSS within one month after sleeve gastrectomy
* Severe medical comorbidities precluding endoscopy or surgery, or limiting life expectancy to less than 2 years in the judgement of the endoscopist
* Uncontrolled coagulopathy or inability to be off anticoagulation or antiplatelet medication for 1 week prior to and after intervention
* Pregnant or planning to become pregnant during period of study participation
* Patient refuses or is unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical success | 6 months post-procedure
  The rate of clinical success, defined as an improvement in symptoms that allowed the patient to avoid further intervention (outside of the predefined treatment algorithm) with a resumption of adequate oral intake and at least 1-point reduction in the Patient Assessment of upper Gastrointestinal Symptoms (PAGI-SYM) questionnaire, at 6 months following last intervention.

SECONDARY OUTCOMES:
Rate of technical success | Immediately post-procedure
  Defined as the completion of planned procedure.
Procedural success as assessed by the PAGI-SYM score | 8 weeks post-procedure
  Procedural success is defined as a 1-point reduction in PAGI-SYM score at 8 weeks following procedure.
Degree of axial deviation per Endoscopic resolution of GSS-related findings | Up to 6 months post-procedure
  Degree of axial deviation post-treatment measured in degrees.
Degree of luminal narrowing per Endoscopic resolution of GSS-related findings | Up to 6 months post-procedure
  Degree of luminal narrowing post-treatment measured as a ratio of the diameter of the narrowest portion over the widest portion of the sleeve.
Degree of axial deviation per Radiologic resolution of GSS-related findings | Up to 6 months post-procedure
  Degree of axial deviation post-treatment measured categorically as: none, mild, moderate or severe.
Degree of luminal narrowing per Radiologic resolution of GSS-related findings | Up to 6 months post-procedure
  Degree of luminal narrowing post-treatment measured as a ratio of the diameter of the narrowest portion over the widest portion of the sleeve.
Presence of delayed contrast flow per Radiologic resolution of GSS-related findings | Up to 6 months post-procedure
  Presence of delayed contrast flow post-treatment measured as either a yes or no.
Percentage of patients maintained off PPI therapy | Up to 6 months post-procedure
  Percentage of patients maintained off proton pump inhibitor (PPI) therapy.
Time to recurrence of symptoms post-treatment in patients with recurrence | Up to 12months post-procedure
  Measured in days.
Rate of adverse events | Up to 6 months post-procedure
  Rate of adverse events will be determined by assessing the number of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Mouen A Khashab, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgos AM, Csendes A, Braghetto I. Gastric stenosis after laparoscopic sleeve gastrectomy in morbidly obese patients. Obes Surg. 2013 Sep;23(9):1481-6. doi: 10.1007/s11695-013-0963-6. PMID 23604695